CLINICAL TRIAL: NCT02464943
Title: Zenith® Dissection Endovascular System in the Treatment of Patients With Acute, Complicated Type B Aortic Dissections
Brief Title: Zenith® Dissection Endovascular System in the Treatment of Patients With Aortic Dissections
Status: Approved for marketing | Type: Expanded Access
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 11-007-CA; NCT02418611 (obsolete NCT alias)
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Aortic Dissection
Keywords: Aorta; Thoracic; Aortic dissection; Type B; DeBakey type III; Endovascular
MeSH Terms: conditions — Aortic Dissection | interventions — Endovascular Aneurysm Repair

INTERVENTIONS:
Device: Endovascular Treatment (Zenith) — Instead of making a large incision in the chest, the physician makes a small incision near each hip to insert, and guides the study device(s) into place in the aorta.
  Other Names: Endovascular graft; Endovascular stent; Stent-graft

SUMMARY:
The Zenith® Dissection extended study is to collect confirmatory safety and effectiveness data on the Zenith® Dissection Endovascular System in the treatment of acute, complicate Type B aortic dissection.

ELIGIBILITY:
Exclusion Criteria:

* < 18 years of age
* Other medical condition(e.g., cancer, congestive heart failure) that may cause the patient to be non-compliant with the protocol, confound the results, or is associated with limited life expectancy (i.e., < 2 years)
* Pregnant, breast-feeding, or planning on becoming pregnant within 60 months
* Unwilling to unable to comply with the follow-up schedule
* Inability or refusal to give informed consent
* Simultaneously participating in another investigative device or drug study. (The patient must have completed the primary endpoint of any previous study at least 30 days prior to enrollment in this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cooper University Hospital, Camden, New Jersey
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia Medical Center, Charlottesville, Virginia